CLINICAL TRIAL: NCT02892110
Title: Advancing Varenicline as a Treatment for Cannabis Use Disorder
Brief Title: Varenicline Treatment for Cannabis Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Aimee McRae-Clark, Professor of Psychiatry, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00058198; UG3DA043231 (NIH)
Record Dates: First submitted 2016-08-30; First posted 2016-09-08 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-10

CONDITIONS: Substance Use Disorder
Keywords: Marijuana use; Varenicline/Chantix; Motivational enhancement therapy
MeSH Terms: conditions — Substance-Related Disorders; Marijuana Use | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Varenicline (Experimental): 2 mg daily
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): 2 mg daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — 2 mg daily
  Other Names: Chantix
  Arms: Varenicline
Drug: Placebo — 2 mg daily
  Arms: Placebo

SUMMARY:
Marijuana is the most commonly used illicit drug. There is high demand for effective interventions for cannabis use disorder, yet few specific treatments for have been developed. This study will evaluate the efficacy of varenicline for reducing marijuana use in people who use marijuana frequently.

ELIGIBILITY:
General Inclusion Criteria

* Must meet DSM-5 criteria for cannabis use disorder and use cannabis at least 3 days per week in the last 30 days.
* Must be between the ages of 18 and 65 years.
* If female and of childbearing potential, must agree to use acceptable methods of birth control for the duration of the trial.
* Must consent to random assignment, and be willing to commit to medication ingestion.
* Must be able to read and provide informed consent.
* Must have body weight >110lbs (50kg) and have BMI between 18 and 35kg/m2
* Must function at an intellectual level and have knowledge of the English language to sufficiently allow for accurate completion of assessments.

Additional Inclusion Criteria for fMRI Eligibility

• Must be right-handed.

General Exclusion Criteria

* Women who are pregnant, nursing, or plan to become pregnant during the course of the study.
* Individuals with severe renal impairment (creatinine clearance less than 30 mL per minute).
* Lifetime history of DSM-5 Bipolar I or II Disorder, Schizophrenia or other psychotic disorder. Stably treated MDD, Dysthymia, GAD, Social Phobia, and Specific Phobia diagnoses are acceptable (i.e. same dose of medication has been prescribed for at least 2 months prior to screening and no changes in current medication expected during course of the trial).
* Suicidal ideation or behavior within the past 6 months. Subjects who are believed to be at suicidal or homicidal risk (answers 'yes' on questions 4 or 5 of C-SSRS) will be referred for assessment by a qualified mental health professional.
* Concomitant use of psychotropic medications, with the exception of stable doses (defined as no dosing adjustments in the past two months) of non-MAO-I antidepressants, non-benzodiazepine anxiolytics, and ADHD medications.
* Current use of medications prescribed for mania or psychosis.
* Current use of buproprion or nortryptiline.
* Moderate or severe non-cannabis substance use disorders within the past 60 days with the exception of tobacco use disorder.
* Individuals taking an investigational agent within the last 30 days before baseline visit.
* Individuals with clinically significant medical disorders or lab abnormalities.
* Any individual at screening with SGOT (AST) or SGPT (ALT) greater than 3 times the upper limit of normal and/or total bilirubin greater than two times the upper limit of normal.
* Individuals with clinically significant cardiovascular disease in the past 6 months (e.g., myocardial infarction, CABG, PTCA, severe or unstable angina, serious arrhythmia, or any clinically significant ECG conduction abnormality.
* Individuals with clinically significant cerebrovascular disease in the past 6 months such as TIA, CVA, or stroke.
* Hypersensitivity to varenicline.
* Individuals who have participated in the clinical trial of any investigative compound within the last 60 days.

Additional Exclusion Criteria for fMRI Eligibility

* Any psychiatric or medical issues, including claustrophobia, ferrous metal implants, pacemakers, or other electronic devices that would interfere with ability to participate in and successfully complete scanning procedures.
* Any person unable to lie still within the fMRI scanner for the required period of time to obtain useful images (use of anxiolytics will not be permitted for anxiety/claustrophobia related to scanning procedures).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee McRae-Clark, PharmD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 35 | 37
Completed | 22 | 25
Not Completed | 13 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 35 | 37 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 37 | 72
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 22 | 27 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 34 | 34 | 68
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 13 | 29
  White | 19 | 23 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 35 | 37 | 72

OUTCOME MEASURES:

1. Primary Outcome: Cannabis Withdrawal Symptoms During Active Treatment
Description: For this outcome, the negative affect subscale items of The Cannabis Withdrawal Scale (items 5 ["I felt nervous], 6 ["I had some angry outbursts"], 7 ["I had mood swings"], 8 ["I felt depressed"], 9 ["I was easily irritated"], 15 ["Life seemed an uphill struggle"], 18 ["I felt physically tense"], restlessness (item 11, "I felt restless), and/or urge to smoke (items 1 and 10, "The only thing I could think about was smoking some cannabis" and "I had been imagining being stoned") were averaged at Weeks 4, 5, and 6 and for an overall 4-6 week value, with minimum score of the subscale being 0 and maximum score being 100 (higher score indicating worse outcome).
Time Frame: 3 weeks (Week 4-6 of active treatment period)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 22 | 25
score on a scale
  Overall Week 4-6 average | 2.23 (4.65) | 3.94 (6.23)
  Week 4 | 2.59 (6.73) | 4.07 (5.81)
  Week 5 | 2.15 (4.84) | 4.27 (7.11)
  Week 6 | 1.96 (4.65) | 3.47 (6.07)

2. Secondary Outcome: Number of Participants With Cannabis Abstinence
Description: Self reported abstinence from Timeline Followback, verified by urine cannabinoid measures
Time Frame: 3 weeks (Week 4-6 of active treatment period)
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 22 | 25
Participants
  Week 4 | 5 | 3
  Week 5 | 4 | 2
  Week 6 | 6 | 2

3. Secondary Outcome: Cannabis Use Quantity
Description: Cannabis use sessions per day measured by Timeline Followback (self-report) at twice weekly visits during Weeks 4, 5 and 6 of the active treatment phase.
Time Frame: 3 weeks (Week 4-6 of active treatment period)
Measure: Mean (95% Confidence Interval); unit: sessions per day
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 22 | 25
sessions per day
  Week 4 | 0.93 [0.54 to 1.33] | 1.33 [0.96 to 1.70]
  Week 5 | 0.89 [0.5 to 1.28] | 1.19 [0.82 to 1.56]
  Week 6 | 0.89 [0.5 to 1.29] | 1.21 [0.84 to 1.58]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from time of consent through last study visit (approximately 8 weeks).
Arm/Group | Varenicline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/37
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/37
Other Adverse Events (participants affected / at risk) | 30/35 | 32/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=35) | Placebo (N=37)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=35) | Placebo (N=37)
Allergies (General disorders) | 1 (1) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Dream disturbance (General disorders) | 15 (15) | 7 (8)
Fatigue (Gastrointestinal disorders) | 4 (4) | 1 (1)
Headache (General disorders) | 9 (11) | 12 (15)
Insomnia (General disorders) | 8 (8) | 9 (10)
Irritability (General disorders) | 2 (2) | 8 (9)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 16 (19) | 9 (10)
URI/cold symptoms (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 7 (11)
Vomiting (Gastrointestinal disorders) | 6 (7) | 5 (7)
Other GI (Gastrointestinal disorders) | 8 (9) | 9 (10)
Dizziness (General disorders) | 3 (4) | 1 (1)

LIMITATIONS AND CAVEATS:
Intended as a proof of concept study; fully powered clinical trials are needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT02892110/Prot_SAP_000.pdf